CLINICAL TRIAL: NCT00681135
Title: Mechanical Plaque Control and Gingivitis Reduction in Fixed Appliance Patients: Comparison of Different Toothbrushing Protocols
Brief Title: Mechanical Plaque Control and Gingivitis Reduction in Fixed Appliance Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sebastian Zingler (Other)
Responsible Party: Sponsor-Investigator, Sebastian Zingler, Dr. med. dent. Sebastian Zingler, University of Jena
Organization: University of Jena (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZKL-08-MHW
Record Dates: First submitted 2008-05-16; First posted 2008-05-21 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Dental Plaque; Gingivitis
Keywords: orthodontics; toothbrush; interdental brush; oral hygiene
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Device: sonic toothbrush (Philips Sonicare® FlexCare, Typ HX6942/04)
- 2 (Experimental)
  Interventions: Device: manual toothbrush / interdental toothbrush (elmex® Inter X medium toothbrush / interdental brush Curaprox®)
- 3 (Experimental)
  Interventions: Device: manual toothbrush (elmex® Inter X medium toothbrush)
- 4 (Active Comparator)
  Interventions: Device: manual toothbrush (elmex® Inter X medium toothbrush)

INTERVENTIONS:
Device: sonic toothbrush (Philips Sonicare® FlexCare, Typ HX6942/04) — toothbrushing with a sonic toothbrush and sealant coating (ProSeal™) of the enemal surface around the brackets
  Other Names: Philips Sonicare® FlexCare
  Arms: 1
Device: manual toothbrush / interdental toothbrush (elmex® Inter X medium toothbrush / interdental brush Curaprox®) — toothbrushing with a manual toothbrush and interdental brush and sealant coating (ProSeal™) of the enemal surface around the brackets
  Other Names: elmex® Inter X medium toothbrush / interdental brush Curaprox®
  Arms: 2
Device: manual toothbrush (elmex® Inter X medium toothbrush) — toothbrushing with a manual toothbrush and sealant coating (ProSeal™) of the enemal surface around the brackets
  Other Names: elmex® Inter X medium toothbrush
  Arms: 3
Device: manual toothbrush (elmex® Inter X medium toothbrush) — toothbrushing with a manual toothbrush without sealant coating of the enemal surface around the brackets
  Other Names: elmex® Inter X medium toothbrush
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether the use of a sonic toothbrush alone is more effective than two other toothbrushing protocols on dental plaque elimination in patients with fixed orthodontic appliances.

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases
* orthodontic appliance (min. 10 completely erupted permanent teeth with brackets/bands)
* informed consent

Exclusion Criteria:

* presence of caries lesion
* antibiotic therapy within the previous 6 months
* diagnosis of early onset periodontitis

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Plaque Indices | every 4 weeks for 3 months
Gingival Indices | every 4 weeks for 3 months

SECONDARY OUTCOMES:
Periodontal parameters | every 4 weeks
Microbiological parameters | every 4 weeks
Molecularbiological parameters | every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. Lux, Professor, Study Chair — Department of Orthodontics, University of Heidelberg
Locations (1):
- Department of Orthodontics, Heidelberg, Baden-Wurttemberg, Germany